CLINICAL TRIAL: NCT00887718
Title: Positron Emission Tomography for Staging, and Treatment Assessment of Response in Lymphomas (the Pet-star Lymphoma Study)
Brief Title: Positron Emission Tomography(PET) in Lymphoma Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 07-0235-C
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Hodgkin's Lymphoma; Non Hodgkin's Lymphoma
Keywords: PET scan and Hodgkin's Lymphoma; PET scan and Non Hodgkin's Lymphoma; PET scan
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET scan for lymphoma assessment (Experimental)
  Interventions: Biological: PET Scan

INTERVENTIONS:
Biological: PET Scan — 18F-Fluorodeoxyglucose (FDG) injection

SUMMARY:
This study examines the role of a diagnostic test called Positron Emission Tomography (PET) scanning in patients with malignant lymphoma. The primary goal of this study is to find out how well PET scanning can detect malignant (cancerous) lymphoma, and how often this extra information will result in a change of stage of disease, or will result in a change in treatment management plans of patients with lymphoma.

DETAILED DESCRIPTION:
It is currently unknown whether modifying treatment based on FDG-PET results is appropriate. However, clinicians are increasingly using the FDG-PET result, where obtained, in deciding management. Consequently, it would be premature to mandate PET-based treatment modifications in this protocol. Patients will be treated with existing protocols at the discretion of their treating oncologists, based on available information. Oncologists will be surveyed as to whether FDG-PET scan results could have (or affect patient management, and the intervention will be recorded).

ELIGIBILITY:
Group A: Newly Diagnosed

Inclusion Criteria:

* Patients > 18 years of age.
* Confirmed diagnosis of HL or NHL (any histology).
* Any Ann Arbor stage.
* Pre-treatment staging including CT of head and neck, chest, abdomen and pelvis, where there is a minimum one equivocal finding on the scan, affecting the assignment of stage or IPI factor (i.e. stage III/IV vs. stage I/II, or a question of extranodal involvement by disease).

Group B: Response Assessment

Inclusion Criteria:

* Patients > 18 years of age.
* Confirmed diagnosis of HL or NHL (any histology).
* Any Ann Arbor stage.
* Pre-treatment staging including CT neck, chest, abdomen and pelvis. If alternate assessment of the neck done by clinical palpitation, ultrasound, or MRI is negative, CT neck is not mandatory.
* Post-treatment staging including CT of head and neck, chest, abdomen and pelvis, at 1 - 6 weeks post-therapy.
* Treated with anthracycline-based chemotherapy, with or without radiation therapy (based on the stage of the disease). For Stage III/IV patients, PET will be done following completion of primary chemotherapy. For stage I/II patients, PET will be done after combined modality therapy, or after chemotherapy alone if this was the primary intention of therapy.
* Patients with residual mass on CT following primary chemotherapy with either "unconfirmed" CR (>75% decrease in size) or PR (³50% decrease in size), based on International workshop criteria.

Exclusion Criteria: Response Assessment

* None Curative treatment Intent
* After initial therapy the response status is: complete response, stable disease, or progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine:the frequency in which the FDG-PET scan result will change the clinical management of the patient, and to record the intervention instituted within 3 months of the PET scan 2)early relapse rates for PET positive, and PET negative patients. | 24 months

SECONDARY OUTCOMES:
To:1) describe & quantify potential changes in clinical practice caused by the adoption of FDG-PET scanning 2)correlate FDG-PET scan findings with disease characteristics, traditional standard response criteria, biopsy results, & early clinical outcome. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Tsang, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada